CLINICAL TRIAL: NCT04557033
Title: My Mindful Moments: A Mindfulness Meditation and Digital Art Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Theresa Jabaley, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-420
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Mindfulness; Meditation
Keywords: Mindfulness; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful Meditation (Experimental): * The activity will include a guided mindfulness meditation and the creation of a digital image on an iPad.
  * The My Moments® application (app) is a tool used to facilitate expressive art creation in a digital photography media
  * Participants will be asked to complete brief surveys before and after the intervention activity.
  Interventions: Other: Mindfulness intervention

INTERVENTIONS:
Other: Mindfulness intervention — My Moments® application (app) is a tool used to facilitate expressive art creation in a digital photography media

SUMMARY:
The purpose of this evidence-based practice project is to evaluate the feasibility of providing a relaxation mindfulness meditation and an expressive digital arts activity among clinical staff at Dana Farber Cancer Institute .

DETAILED DESCRIPTION:
This project provides an opportunity for patient care staff in an ambulatory oncology setting to participate in and evaluate an activity that includes a mindfulness meditation technique and an expressive digital arts activity.

This study will be conducted to evaluate the feasibility of providing a mindfulness meditation and digital imagery activity.

* The activity will include a guided mindfulness meditation and the creation of a digital image on an iPad.
* Participants will be asked to complete brief surveys before and after the intervention activity.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Currently employed at Dana Farber Cancer Institute
* Providing patient care on Yawkey

Exclusion Criteria:

* Not an employee of Dana Farber Cancer Institute
* Not providing Patient Care on Yawkey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participation-Feasibility | 1 year
  ≥50% of staff choose to participate=Feasibility. This measure of feasibility will be evaluated by calculating index scores of the percentage of clinical staff who choose to participate
Percentage Completion of Full Activity-Feasibility | 1 year
  > 80% of those who participate complete the activity=Feasibility. This measure of feasibility will be evaluated by index scores of the percentage of clinical staff who complete the full activity
Mean Completion Time-Feasibility | 1 year
  The activity is completed by the group in 40 minutes or less-Feasibility. This measure of feasibility will be evaluatedby individual group completions times and overall analysis of descriptive statistics on the time for completion of the activity by all groups.

SECONDARY OUTCOMES:
Change in Anxiety Score | 1 Year
  Changes in participant state anxiety will be evaluated using the visual analogue scale in measuring state anxiety. The electronic scale displays a horizontal line divided into 30 equal-sized partitions. The left edge of the scale is marked "calm" and the right edge is marked "anxious." A sliding locator is positioned at the midpoint of the scale. The participant is instructed to use the computer mouse to place the locator at the scale position representing their current level of anxiety. The score is automatically calculated by rounding the relative distance of the locator from the left edge of the scale to the nearest integer value between 0 and 30. A higher score indicates greater anxiety. A comparison of scores pre- and post- intervention by calculating a paired t-test comparison of means

CONTACTS AND LOCATIONS:
Overall Officials: Terri Jabaley, Ph.D, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

DOCUMENTS (1):
  • Study Protocol (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT04557033/Prot_000.pdf